CLINICAL TRIAL: NCT02745184
Title: Clinical Efficacy and Safety of Autologous Lung Stem Cell Transplantation in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Regend Therapeutics (Industry)
Responsible Party: Principal Investigator, Wei Zuo, Professor, Shanghai East Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201602101
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung stem cells (Experimental): Patients will receive 0.5-5x10^6 (0.5-5 million)/Kg/person cells of clinical grade lung stem cells (LSCs)injected via fiberoptic bronchoscopy after fully lavage of the localized lesions.
  Interventions: Biological: Lung stem cells

INTERVENTIONS:
Biological: Lung stem cells — Patients will receive 0.5-5x10^6 (0.5-5 million) /Kg/person cells of clinical grade lung stem cells (LSCs) injected via fiberoptic bronchoscopy after fully lavage of the localized lesions.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic and ultimately fatal disease characterized by a progressive damage of lung structure and decline in lung function.This study intends to carry out an open, single-center, non-randomized, self control phase I clinical trial. During the treatment, lung stem cells will be isolated from patients' own bronchi and expanded in vitro. Cultured cells will be injected directly into the lesion by fiberoptic bronchoscopy after lavage. After 24-week observation, the investigators will evaluate the safety and efficacy of the treatment by measuring the key clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 50 to 75;
2. Subjects diagnosed with IPF according to guidelines for the diagnosis of idiopathic pulmonary fibrosis 2018 edition;
3. Subjects with 30%~79% of the predicted value in diffusing capacity for carbon monoxide (DLCO) in pulmonary function tests 3 months before screening;
4. Subjects with typical High-resolution computed tomography (HR-CT) imaging findings of idiopathic pulmonary fibrosis in the past 12 months;
5. Subjects tolerant to bronchofiberscope;
6. Subjects fully informed of the purpose, method and possible discomfort of the trial, agreeing to participate in the test, and voluntarily signing the informed consent;
7. Subjects with good adherence, willingness to take medication and regular follow-up examinations as required by the protocol;
8. Subjects able to understand and cooperate with the completion of pulmonary function tests.

Exclusion Criteria:

1. Subjects who cannot tolerate cell therapy;
2. Pregnant or lactating women;
3. Subjects with syphilis or any of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) positive antibody; Of which stable HBV carriers after drug treatment (DNA titer ≤500 IU/mL or copy number <1000 copies/mL) and cured hepatitis C patients (HCV RNA is negative) can be enrolled;
4. Subjects with malignant tumors or a history of malignant tumors;
5. Subjects with serious significant pulmonary infection and needing anti-infection treatment;
6. Subjects with taking drugs which caused lung fibroblast such as amiodarone in a long term before screening;
7. Subjects with infections in lung or other site, including bacterial and viral infections, requiring intravenous treatment before cell transplantation;
8. Subjects with a history of invasive or noninvasive mechanical ventilation within 4 weeks;
9. Subjects with any of the following lung diseases: asthma, active tuberculosis, pulmonary embolism, pneumothorax, pulmonary hypertension, pneumoconiosis, etc.; lung cancer, bronchiolitis obliterans or other active lung disease; Pneumonia currently or within the last 4 weeks; Pneumonectomy Previously;
10. Subjects needing oxygen therapy currently (oxygen therapy time> 15h/d);
11. Subjects suffering from serious other systemic diseases, such as myocardial infarction, unstable angina, liver cirrhosis, acute glomerulonephritis, connective tissue disease, etc.;
12. Subjects with following results : leukopenia (leukopenia < 4×10^9/L) or agranulocytosis (leukocyte < 1.5×10^9/L or neutrophils < 0.5×10^9/L) of any cause; Blood creatinine > 2.5 times the upper limit of normal; Alanine transaminase (ALT) and Aspartate transaminase (AST) > 2.5 times the upper limit of normal values in the laboratory tests;
13. Subjects with a history of mental illness or suicide risk, epilepsy or other central nervous system disorders;
14. Subjects with severe arrhythmias (such as ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or atrioventricular block of degree II or above, shown by 12-lead Electrocardiogram (ECG);
15. Subjects with a history of abusing alcohol and illicit drug;
16. Subjects with serious heart disease [New York Heart Association (NYHA) class III-IV];
17. Subjects who are allergic to cattle products;
18. Subjects who participated in other clinical trials in the past 3 months;
19. Subjects with poor compliance and difficult to complete the investigation;
20. Investigators, employees of research centers or family members of them (none of whom are suitable to participate in the trial to ensure the objectivity of the research);
21. Subjects who had an acute exacerbation of IPF or hospitalized for other respiratory diseases 3 or more times in the past 1 year;
22. Subjects who take nintedanib for medication within 1 month, or plan to continue taking nintedanib for medication;
23. Subjects with other acquired or congenital immunodeficiency disorders, or with a history of organ transplantation or cell transplant therapy;
24. Subjects whose expected survival may be less than one year judged by the investigator;
25. Male participants of childbearing potential and female participants within childbearing age were reluctant to use effective contraception from the time of signing the informed consent to 6 months after cell therapy;
26. Subjects assessed as inappropriate to participate in this clinical trial by investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was the incidence and severity of the cell therapy-related AEs | 24 weeks
  To evaluate the safety of the drugs

SECONDARY OUTCOMES:
Incidence of complication related to bronchoscopy | 1 week
Evaluation of cell therapy efficacy through DLCO-SB test | 24 weeks
exercise tolerance test (6MWD) | 24 weeks
Life quality: assessed by St. George respiratory questionnaire (SGRQ) | 24 weeks
Change from baseline in forced vital capacity (FVC) | 24 weeks
  FVC indicates the volume of air that can forcibly be blown out after full inspiration.
Change from baseline in imaging of lung by high resolution computed tomography (HR-CT) | 24 weeks
  Images of lung will be analyzed to indicate the newly-derived pulmonary structure
IPF exacerbation events | 24 weeks
Change from baseline in forced expiratory volume in one second (FEV1) | 24 weeks
  FEV1 is the volume of breath exhaled with effort in one second.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540